CLINICAL TRIAL: NCT05292664
Title: A Phase I Study of Venetoclax in Combination With Cytotoxic Chemotherapy, Including Calaspargase Pegol, for Children, Adolescents and Young Adults With High-Risk Hematologic Malignancies
Brief Title: Venetoclax Basket Trial for High Risk Hematologic Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Andrew E. Place, MD (Other)
Collaborators: AbbVie (Industry); Servier (Industry); Children's Cancer Research Fund (Other); University of Colorado, Denver (Other); Boston Children's Hospital (Other); Gateway for Cancer Research (Other)
Responsible Party: Sponsor-Investigator, Andrew E. Place, MD, Sponsor-Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-757
Record Dates: First submitted 2022-03-05; First posted 2022-03-23 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Myelodysplastic Syndromes, de Novo; Myelodysplastic Syndromes, Secondary; Myelodysplastic Syndromes, Previously Treated; Treatment-Related Acute Myeloid Leukemia; Therapy-Related Myelodysplastic Syndrome; Acute Lymphoblastic Leukemia, in Relapse; Acute Lymphoblastic Leukemia With Failed Remission; Lymphoblastic Lymphoma, in Relapse; Lymphoblastic Lymphoma, Refractory; Acute Leukemia of Ambiguous Lineage in Relapse; Acute Leukemia of Ambiguous Lineage
Keywords: Myelodysplastic Syndrome (MDS); Treatment-related Acute Myelogenous Leukemia; AML arising from MDS; Relapsed or Refractory Acute Lymphoblastic Leukemia; Relapsed or Refractory Acute Lymphoblastic Lymphoma; Relapsed or Refractory MDS; Treatment-related MDS; Relapsed or Refractory Acute leukemia of ambiguous lineage
MeSH Terms: conditions — Myelodysplastic Syndromes; Neoplasm Metastasis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute; Recurrence | interventions — venetoclax; Azacitidine; Cytarabine; Methotrexate; Hydrocortisone; Cortisone; hydrocortisone sodium phosphate; Leucovorin; Dexamethasone; dexamethasone 21-phosphate; dexamethasone acetate; Vincristine; Doxorubicin; Dexrazoxane; calaspargase pegol; asparaginase erwinia chrysanthemi recombinant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): For Part 1, participants will receive:
  * Patients with myelodysplastic syndrome (MDS) or acute myelogenous leukemia (AML). It is expected that up to 18 people will participate in Part 1 (Dose Determination) and an additional 14-20 people will participate in Part 2 (Dose Expansion) of this cohort Treatment cycle is approximately 28 days for up to 4 cycles
    * Venetoclax-once daily on predetermined days per protocol
  * Azacitidine-once daily on predetermined days per protocol
    * Cytarabine, Methotrexate, Hydrocortisone and Leucovorin will be given only if MDS/leukemia cells are detected in spinal fluid per determination of treating physician
  Interventions: Drug: Venetoclax; Drug: Azacitidine; Drug: Cytarabine; Drug: Methotrexate; Drug: Hydrocortisone; Drug: Leucovorin
- Cohort B (Experimental): Patients with myelodysplastic syndrome (MDS) or acute myelogenous leukemia (AML) with an underlying genetic condition that increases their risk for developing treatment-related toxicities. It is expected that up to 18 people will participate in Part 1 (Dose Determination) and an additional 6 people will participate in Part 2 (Dose Expansion) of this cohort.
  * Venetoclax-once daily on predetermined days per protocol
  * Azacitidine-once daily on predetermined days per protocol
  * Cytarabine, Methotrexate, Hydrocortisone and Leucovorin will be given only if MDS/leukemia cells are detected in spinal fluid per determination of treating physician
  Interventions: Drug: Venetoclax; Drug: Azacitidine; Drug: Cytarabine; Drug: Methotrexate; Drug: Hydrocortisone; Drug: Leucovorin
- Cohort C (Experimental): Patients with relapsed/refractory acute lymphoblastic leukemia (ALL), lymphoblastic lymphoma (LBL) or acute leuekmai of ambiguous lineage. It is expected that up to 18 people will participate in Part 1 (Dose Determination) and an additional 12 people will participate in Part 2 (Dose Expansion) of this cohort.
  Cohort C: Treatment cycle is approximately 32 days for one cycle and will be a single treatment cycle:
  Dosage, duration and timings as outlined in protocol.
  * Venetoclax
  * Dexamethasone
  * Vincristine
  * Doxorubicin
  * Dexrazoxane
  * Calaspargase pegol
    ---Short acting Erwinia preparations (recombinant or native Erwinia asparaginase) may be used for participants with known pegaspargase or calaspargase pegol allergy
  * Cytarabine
  * Methotrexate
  * Hydrocortisone
  * Leucovorin- *Cytarabine, Methotrexate, Hydrocortisone and Leucovorin may be given more frequently if leukemia/lymphoma cells are detected in spinal fluid),
  Interventions: Drug: Venetoclax; Drug: Cytarabine; Drug: Methotrexate; Drug: Hydrocortisone; Drug: Leucovorin; Drug: Dexamethasone; Drug: Vincristine; Drug: Doxorubicin; Drug: Dexrazoxane; Drug: Calaspargase Pegol; Drug: Erwinia asparaginase

INTERVENTIONS:
Drug: Venetoclax — Tablet taken orally
  Other Names: Venclexta
Drug: Azacitidine — Taken intravenously
  Other Names: Vidaza
  Arms: Cohort A; Cohort B
Drug: Cytarabine — Lumbar Puncture
  Other Names: Ara-C; Arabinosylcytosine
Drug: Methotrexate — Lumbar Puncture
  Other Names: Amethopterin; Methotrexate Sodium; MTX
Drug: Hydrocortisone — Lumbar Puncture
  Other Names: Cortisone; Hydrocortisone Sodium Succinate; Hydrocortisone Sodium Phosphate
Drug: Leucovorin — Taken Orally or intravenously
  Other Names: Calcium Leucovorin,; Citrovorum Factor; Folinic Acid
Drug: Dexamethasone — Taken Orally or intravenously
  Other Names: dexamethasone sodium phosphate; dexamethasone acetate
  Arms: Cohort C
Drug: Vincristine — Taken intravenously
  Other Names: Vincristine Sulfate; LCR; VCR
  Arms: Cohort C
Drug: Doxorubicin — Taken intravenously
  Other Names: Adriamycin; Rubex
  Arms: Cohort C
Drug: Dexrazoxane — Taken intravenously
  Other Names: Zinecard
  Arms: Cohort C
Drug: Calaspargase Pegol — Taken intravenously
  Other Names: Asparlas
  Arms: Cohort C
Drug: Erwinia asparaginase — Given as intramuscular injection
  Other Names: Rylze or native Erwinia asparaginase
  Arms: Cohort C

SUMMARY:
This trial is evaluating the safety and tolerability of venetoclax with chemotherapy in pediatric and young adult patients with hematologic malignancies, including myelodysplastic syndrome (MDS), acute myeloid leukemia derived from myelodysplastic syndrome (MDS/AML), and acute lymphoblastic leukemia (ALL)/lymphoblastic lymphoma (LBL).

The names of the study drugs involved in this study are below. Please note this is a list for the study as a whole, participants will receive drugs according to disease cohort.

* Venetoclax
* Azacitidine
* Cytarabine
* Methotrexate
* Hydrocortisone
* Leucovorin
* Dexamethasone
* Vincristine
* Doxorubicin
* Dexrazoxane
* Calaspargase pegol
* Hydrocortisone

DETAILED DESCRIPTION:
This is an investigator-initiated open-label multi-institutional phase I study of venetoclax combination therapy in both myeloid and lymphoid hematologic malignancies. This study is designed as a basket trial with three separate cohorts. All cohorts include a dose finding portion (Part I) followed by a dose expansion at the Recommended Phase II dose (RP2D, Part II).

This research study is looking to learn more about how Venetoclax works and aims to determine the safest, highest possible dose that can be combined with standard of care chemotherapies. Because of this, not everyone who participates in this research study may receive the same dose of the study drug. The dose participants receive will depend on the number of participants who have been enrolled in the study previously and how well the doses have been tolerated.

Study procedures include screening for eligibility as well as study treatment visits including evaluations and follow up visits.

* Cohort A: Patients with myelodysplastic syndrome (MDS), acute myelogenous leukemia arising from MDS (MDS/AML) or treatment-related myeloid neoplasms (tMDS/AML). It is expected that up to 18 people will participate in Part 1 (Dose Determination) and an additional 14-20 people will participate in Part 2 (Dose Expansion) of this cohort.
* Cohort B: Patients with myelodysplastic syndrome (MDS), acute myelogenous leukemia arising from MDS (MDS/AML) or treatment-related myeloid neoplasms (tMDS/AML) with an underlying genetic condition that increases their risk of experiencing toxic side effects of chemotherapy. It is expected that up to 18 people will participate in Part 1 (Dose Determination) and an additional 6 people will participate in Part 2 (Dose Expansion) of this cohort.
* Cohort C: Patients with relapsed/refractory acute lymphoblastic leukemia (ALL) or lymphoblastic lymphoma (LBL). It is expected that up to 18 people will participate in Part 1 (Dose Determination) and an additional 12 people will participate in Part 2 (Dose Expansion) of this cohort.

This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied. The U.S. Food and Drug Administration (FDA) has not approved Venetoclax for use in children. However, Venetoclax is FDA-approved as a treatment for certain types of leukemia in adults. It is actively being studied in children and adults with other types of cancer. Information from these research studies has suggested that venetoclax may also be effective in treating participants with MDS or leukemia, including MDS or leukemia that did not respond to standard treatment or that has come back after standard treatment. The survival of cancer cells is controlled by proteins within the cancer cell. One of these proteins is called BCL-2. The study drug, venetoclax, blocks this protein and is thought to reduce cell survival in some cancer cells.

ELIGIBILITY:
Inclusion Criteria

Cohort A Inclusion Criteria:

* MDS, AML arising from MDS (MDS/AML), therapy related myeloid neoplasm (tMDS/AML) meeting at least one of the following criteria:

  * MDS with excess blasts (>10%)
  * MDS with blasts <10% with high-risk features
  * MDS refractory to initial treatment
  * Relapsed MDS
  * MDS/AML: May be newly diagnosed or relapsed/refractory disease.
  * Therapy related myeloid neoplasm (tMDS/AML): May be initial or relapsed/refractory disease.

    * Note: MDS or MDS/AML may be derived from a germline predisposition to myeloid malignancy as long as that condition does not confer increased toxicity to treatment.
* Age ≤ 40 years of age, except the following subjects that must be <18 years to enroll

  * Subjects with MDS/AML that have not received prior therapy
  * Subjects enrolled onto Dose level -2.
* Lansky/Karnofsky performance status ≥ 50%
* Participants must have fully recovered from the acute toxic effects of all and meet all of the following criteria:

  * Myelosuppressive chemotherapy: 14 days, or 5 half-lifes (whichever is shorter) must have elapsed since the completion of myelosuppressive therapy. Individuals may have received any of the following medications without a "wash-out" period

    * Standard maintenance therapy: dexamethasone/prednisone, vincristine, 6MP, low dose methotrexate)
    * Hydroxyurea
    * Intrathecal chemotherapy with methotrexate, hydrocortisone and/or cytarabine.
  * Radiation therapy (XRT):

    * Total Body Irradiation (TBI) or cranial radiation therapy: Must have been completed more than 90 days prior to study entry
    * XRT for chloroma does not require a washout period.
    * Palliative XRT does not require a washout
  * Small molecule inhibitors (BCR-ABL or FLT3 inhibitors, for example): 7 days, or 5 half-lifes, whichever is shorter) must have elapsed since the completion of therapy. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur.
  * Immunotherapy: At least 30 days after the administration of any type of immunotherapy, including, but not limited to, tumor vaccines, chimeric antigen receptor (CAR) therapy, other immune effector cell therapy and checkpoint inhibitors.
  * Monoclonal antibodies: At least 3 half-lives of the antibody
  * Prior hematopoietic stem cell transplant (HSCT):

    * Allogeneic HSCT > 90 days of study entry
    * No evidence of graft-versus-host-disease (GVHD)
  * Adequate organ function, as defined by

    * Serum alanine aminotransferase (ALT) ≤5X upper limit of normal (ULN)
    * Direct bilirubin ≤ 3X
    * Ejection fraction ≥ 50% or shortening fraction of ≥ 24% on screening echocardiogram.
  * Female participants of childbearing potential must have a negative urine or serum HCG prior to study entry and at the start of therapy. All females of childbearing potential must refrain from breastfeeding during study participation, and all male and females of childbearing potential must agree to use an effective form of contraception (abstinence, hormonal, or barrier) prior to study entry, for duration of participation, and for a minimum of 30 days following the last dose of treatment.

Cohort B Inclusion Criteria

* MDS, MDS/AML, therapy related myeloid neoplasm (tMDS/AML) that is derived from the following germline disorders:

  * Dyskeratosis Congenita or associated telomeropathies
  * Fanconi Anemia
  * Nijmegen Breakage
  * Other related disorders with high risk of toxicity may be eligible for this cohort after discussion with the Sponsor-Investigator.
* And meets at least one the following disease characteristics:

  * MDS with excess blasts (>10%)
  * MDS with blasts <10% with high-risk features
  * MDS refractory to initial treatment
  * Relapsed MDS
  * MDS/AML: May be newly diagnosed or relapsed/refractory disease.
  * Therapy related myeloid neoplasm (tMDS/AML): May be initial or relapsed/refractory disease.
* Age ≤ 40 years of age
* Lansky/Karnofsky performance status ≥ 50%
* Participants must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study and meet all of the following criteria:

  * Myelosuppressive chemotherapy: 14 days, or 5 half-lifes (which ever is shorter) must have elapsed since the completion of myelosuppressive therapy. Individuals may have received any of the following medications without a "wash-out" period

    * Standard maintenance therapy: dexamethasone/prednisone, vincristine, 6MP, low dose methotrexate
    * Hydroxyurea
    * Intrathecal chemotherapy with methotrexate, hydrocortisone and/or cytarabine.
  * Radiation therapy (XRT):

    * Total Body Irradiation (TBI) or cranial radiation therapy: Must have been completed more than 90 days prior to study entry
    * XRT for chloroma does not require a washout period.
    * Palliative XRT does not require a washout
  * Small molecule inhibitors (BCR-ABL or FLT3 inhibitors, for example): 7 days, or 5 half-lifes, whichever is shorter) must have elapsed since the completion of therapy. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur.
  * Immunotherapy: At least 30 days after the administration of any type of immunotherapy, including, but not limited to, tumor vaccines, chimeric antigen receptor (CAR) therapy, other immune effector cell therapy and checkpoint inhibitors.
  * Monoclonal antibodies: At least 3 half-lives of the antibody
  * Prior hematopoietic stem cell transplant (HSCT): Must meet all of the following conditions:

    * Allogeneic HSCT > 90 days of study entry
    * No evidence of graft-versus-host-disease (GVHD)
* Adequate organ function, as defined by

  * Serum alanine aminotransferase (ALT) ≤5X upper limit of normal (ULN)
  * Direct bilirubin ≤ 3X upper limit of normal for age and institution.
* Ejection fraction ≥ 50% or shortening fraction of ≥ 24% on screening echocardiogram.
* Because of the teratogenic effects of venetoclax on developing fetuses, female participants of childbearing potential must have a negative urine or serum HCG prior to study entry and at the start of therapy. All females of childbearing potential must refrain from breastfeeding during study participation, and all male and females of childbearing potential must agree to use an effective form of contraception (abstinence, hormonal, or barrier) prior to study entry, for duration of participation, and for a minimum of 30 days following the last dose of treatment.

Cohort C Inclusion Criteria

* Part I: B-cell or T-cell acute lymphoblastic leukemia (ALL), mixed phenotype acute lymphoblastic leukemia (MPAL) or lymphoblastic lymphoma (LBL) in first or greater relapse or refractory to at least 1 prior remission induction attempt.

  * For ALL/MPAL: Bone marrow involvement ≥ 5% by aspirate morphology or ≥ 1% assessable by flow cytometry or validated molecular minimal residual disease (MRD) testing
  * For LBL: Radiographically detectable mass or lymph node involvement
* Part II: Histologically confirmed diagnosis of one of the following:

  * T-cell acute lymphoblastic leukemia (T-ALL) or T-cell lymphoblastic lymphoma (T-LBL) in first or greater relapse or refractory to at least 1 prior remission induction attempt.

    * For T-ALL: Bone marrow involvement ≥ 5% by aspirate morphology or ≥ 1% assessable by morphology, flow cytometry or validated MRD testing
    * For T-LBL (biopsy proven at current or prior relapse): Radiographically detectable mass or lymph node involvement OR
  * Relapsed or refractory B-cell acute lymphoblastic leukemia (B-ALL) with bone marrow involvement ≥1% (assessable by morphology, flow cytometry or validated MRD testing) and at least one of the following characteristics:

    * First relapse with adverse biologic determinants as described below:

      * KMT2A rearrangement
      * Low hypodiploidy, defined as ≤ 40 chromosomes
      * t(17;19)
      * IKZF1 deletion (without targetable ABL1 fusion)
      * Ph-like ALL (without targetable ABL1 fusion)
      * Other biologic determinants with adverse prognosis in discussion with the Sponsor-Investigator
    * Early first bone marrow relapse occurring <36 months from initial diagnosis
    * Primary refractory ALL that has failed 1 prior induction attempt
* Age: ≥ 1 and ≤ 21 years of age
* Lansky/Karnofsky performance status ≥ 50%
* Participants must have fully recovered from the acute toxic effects of all prior and meet all of the following criteria:

  * Myelosuppressive chemotherapy: 14 days, or 5 half-lives, whichever is shorter, must have elapsed since the completion of myelosuppressive therapy. Individuals may have received any of the following medications without a "wash-out" period:

    * Standard maintenance therapy: dexamethasone/prednisone, vincristine, 6MP, low dose methotrexate
    * Hydroxyurea
    * Intrathecal chemotherapy with methotrexate, hydrocortisone and/or cytarabine.
  * Radiation therapy (XRT):

    * Total Body Irradiation (TBI) or cranial radiation therapy: Must have been completed more than 90 days prior to study entry
    * XRT for chloroma does not require a washout period.
    * Palliative XRT does not require a washout
  * Small molecule inhibitors (BCR-ABL or FLT3 inhibitors, for example): 7 days, or 5 half-lifes, whichever is shorter) must have elapsed since the completion of therapy. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur.
  * Immunotherapy: At least 30 days after the administration of any type of immunotherapy, including, but not limited to, tumor vaccines, chimeric antigen receptor (CAR) therapy, other immune effector cell therapy and checkpoint inhibitors.
  * Monoclonal antibodies: At least 3 half-lives of the antibody after the last dose of a monoclonal antibody
  * Prior hematopoietic stem cell transplant (HSCT): Patients who have received HSCT are eligible, but must meet all of the following conditions:

    * Allogeneic HSCT > 90 days of study entry
    * No evidence of graft-versus-host-disease (GVHD)
* Adequate organ function, as defined by the following laboratory values:

  * Serum alanine aminotransferase (ALT) ≤5X upper limit of normal (ULN), unless deemed secondary to leukemic involvement in discussion with site PI.)
  * Direct bilirubin ≤ 3X upper limit of normal for age and institution.
  * Serum amylase ≤ 3X institutional ULN .
* Cardiac function as defined as below:

  * Ejection fraction ≥ 50% or shortening fraction of ≥ 24% on screening echocardiogram.
  * Maximum prior cumulative doxorubicin dose ≤ 360 mg/m2 or equivalent
* Because of the teratogenic effects of venetoclax on developing fetuses, female participants of childbearing potential must have a negative urine or serum HCG prior to study entry and at the start of therapy. All females of childbearing potential must refrain from breastfeeding during study participation, and all male and females of childbearing potential must agree to use an effective non-hormonal form of contraception (abstinence, barrier) prior to study entry, for duration of participation, and for a minimum of 3 months following the last dose of treatment (as calaspargase pegol can render hormonal contraceptives ineffective).

Exclusion Criteria

Cohort A Exclusion Criteria

* Use of strong or moderate CYP3A inhibitors/inducers within 3 days of study entry
* Individuals who have had a stem cell transplant and are still receiving treatment for GVHD or GVHD prophylaxis, or who have evidence of acute GVHD
* Individuals with known active hepatitis; baseline testing not required.
* Patients with systemic infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment.
* Patients known to have human immunodeficiency virus (HIV) infection; baseline testing for HIV is not required.
* Pregnant or nursing women are excluded.
* Individuals with significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.

Cohort B Exclusion Criteria

* Use of strong or moderate CYP3A inhibitors/inducers within 3 days of study entry
* Individuals who have had a stem cell transplant and are still receiving treatment for GVHD or GVHD prophylaxis, or who have evidence of acute GVHD
* Individuals with known active hepatitis; baseline testing not required.
* Patients with systemic infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment.
* Patients known to have human immunodeficiency virus (HIV) infection; baseline testing for HIV is not required.
* Pregnant or nursing women are excluded.
* Individuals with significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.

Cohort C Exclusion Criteria

* Use of strong or moderate CYP3A inhibitors/inducers within 3 days of study entry
* Individuals who have had a stem cell transplant and are still receiving treatment for GVHD or GVHD prophylaxis, or who have evidence of acute GVHD, or who are less than 90 days from stem cell infusion
* Individuals with known active hepatitis; baseline testing not required.
* Patients with systemic fungal, bacterial, viral or other infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment.
* Patients known to have human immunodeficiency virus (HIV) infection; baseline testing for HIV is not required.
* Pregnant or nursing women are excluded
* Individuals with significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
* Individuals with a history of allergic reactions to any of the agents being used in this trial, with the exception of pegaspargase or calaspargase pegol. Participants with a history of allergy to pegylated formulation of asparasginase are allowed on study but should receive commercial supply of asparaginase Erwinia chrysanthemi (Erwinaze), crisantaspase (Erwinase), or asparaginase erwinia chrysanthemi (recombinant)-rywn (Rylaze) instead of calaspargase pegol (see Sections 6.2.6 and 6.2.7). Individuals with a history of allergy to Erwinaze, Erwinase or Rylaze are excluded from the study.
* History of asparaginase-associated pancreatitis.
* Known, active and propagating deep venous thrombus (DVT).
* Individuals with isolated CNS or testicular relapse.
* Presence of surface immunoglobulin by flow cytometry and/or known t(8;14), t(2;8), or t(8;22).
* Individuals with a history of a different malignancy are ineligible except for the following circumstances:

  * Individuals are eligible if they have been disease-free for at least 1 year and are deemed by the investigator to be at low risk for recurrence of that malignancy.
  * Individuals with the following cancers are eligible if diagnosed and treated within the past year: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.

Ages: 1 Year to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2026-07-02 (Estimated); Study Completion 2028-07-02 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | MTD determined during first cycle of treatment (Cohorts A&B: max. 35 Days; Cohort C: 32 days)
  To determine the maximum tolerated dose (MTD of venetoclax given in combination with regimen-prescribed chemotherapy. The MTD is defined as the dose level associated with observed DLTs in <33% of enrolled subjects
Recommended Phase II Dose | RP2D is determined during first cycle of treatment (Cohorts A&B: max. 35 Days; Cohort C: 32 days)
  To determine the Recommended Phase 2 Dose (RP2D) of venetoclax given in combination with regimen-prescribed chemotherapy.
  The RP2D is defined either as the MTD or maximum dose tested should MTD not be reached.
Incidence of Grade 2 or Higher Treatment-Related Toxicity | Up to 30 days after last dose of study treatment
  All grade 2 or higher adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAE v5 criteria. Incidence is the number of patients experiencing at least one treatment-related grade 2 or higher AE of any type during the time of observation.
Incidence of calaspargase pegol related toxicities | Cohort C only: Up to 30 days after last dose of study treatment
  Describe the incidence and severity of calaspargase pegol-related toxicities in subjects with relapsed/refractory ALL/LBL per collected Adverse Events using CTCAE v5 criteria.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Cohorts A&B: Best response during up to 4 cycles (each cycle is max 35 days). Cohort C: Response to treatment after 32 days
  ORR will be defined as the number of patient experiencing complete remission (CR), complete remission with incomplete platelet recovery (CRp), complete remission with incomplete count recovery (CRi) and partial response.
Complete Remission (CR) Rate | Cohorts A&B: Best response during up to 4 cycles (each cycle is max 35 days). Cohort C: Response to treatment after 32 days
  CR Rate is defined as the percentage of participants that reach Complete Remission (CR):
  Cohorts A and B:
  * Bone marrow < 5% myeloblasts by flow cytometry.
  * No evidence of circulating blasts or extramedullary disease AND
  * Platelet count ≥50k/uL (or to pre-treatment baseline) and transfusion independent for 7 days AND
  * Neutrophil count ≥500 cells/uL without G-CSF support.
  Cohort C (Leukemia):
  * Absolute phagocyte count (APC) ≥1000/μL and platelets ≥75,000/μL without transfusions and/or exogenous growth factor support AND
  * Bone marrow with evidence of trilineage hematopoiesis and with <5% blasts AND
  * No evidence of extramedullary disease
Complete Remission with Inadequate Count Recovery (CRi) Rate | Cohort C: Response to treatment
  Cohort C only:
  * APC <1000/μL and/or platelets <75,000/μL AND
  * Bone marrow with <5% blasts AND
  * No evidence of extramedullary disease
Complete Remission with Inadequate Platelet Recovery (CRp) Rate | Cohorts A&B: Best response during up to 4 cycles (each cycle is max 35 days). Cohort C: Response to treatment after 32 days
  CRp Rate is defined as the percentage of participant that reach to CRp:
  Cohorts A &B:
  * A bone marrow with <5% blasts AND
  * No evidence of circulating blasts or extramedullary disease AND
  * Recovery of absolute neutrophil counts (ANC > 500/μL), but with insufficient recovery of platelets (PLT counts <50,000 ul), and platelet transfusion independence (defined as no platelet transfusion x 1 week)
  Cohort C:
  * Absolute neutrophil count (APC ≥1000/μL) AND
  * Platelets < 75,000/μL AND
  * Bone marrow with evidence of trilineage hematopoiesis and with <5% blasts AND
  * No evidence of extramedullary disease
2-year Overall Survival (OS) | Up to 2 years
  Based on the Kaplan-Meier method defined as the time from study entry to death or censored at date last known alive
2-year Event free survival (EFS) | Up to 2 years
  EFS is defined as the time from first dose of study treatment until evidence of progression to leukemia, relapse of MDS or leukemia after HSCT, or death from any cause.

OTHER OUTCOMES:
Proportion of patients to receive all doses of venetoclax | Determined during first cycle of treatment (Cohorts A&B: max. 35 Days, Cohort C: 32 days)
  Estimate the proportion of patients who are able to receive all doses of venetoclax in cycle 1 for each cohort.
Percentage of patients to proceed to Hematopoietic Stem Cell Transplant (HSCT) | Up to 2 years
  Define the percentage of patients in cohorts A&B who successfully proceed to HSCT after treatment with venetoclax combination therapy

CONTACTS AND LOCATIONS:
Overall Officials: Andrew E Place, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - University of California San Francisco-Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta at Arthur M. Blank Hospital, Atlanta, Georgia
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Andrew E. Place (Sponsor-Investigator). The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu